CLINICAL TRIAL: NCT04453085
Title: An Extension Study of JR-171-101 Study in Patients With Mucopolysaccharidosis Type I
Brief Title: An Extension Study of JR-171-101 Study in Patients With Mucopolysaccharidosis Type I (MPS I)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-171-102
Record Dates: First submitted 2020-06-04; First posted 2020-07-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis I
Keywords: Mucopolysaccharidosis I
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose level 1 (Experimental): 2.0 mg/kg/week
  Interventions: Drug: JR-171
- Dose level 2 (Experimental): 4.0 mg/kg/week
  Interventions: Drug: JR-171

INTERVENTIONS:
Drug: JR-171 — Intravenous (IV) infusion
  Other Names: lepunafusp alfa

SUMMARY:
Phase I/II, open label, multicenter, multinational (Japan, Brazil and the US) extension study of JR-171-101 (NCT04227600) for the treatment of MPS I

DETAILED DESCRIPTION:
Patients who have completed the Part2 of JR-171-101 study (NCT04227600) and fulfill all eligibility criteria can be enrolled in this JR-171-102 study. In the JR-171-102 study, subjects will receive either 2.0 or 4.0 mg/kg/week of JR-171 intravenously at the same doses received at Week 12 of the JR-171-101 study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the Part 2 of JR-171-101 study
* A patient from whom written informed consent can be obtained. If the patient is aged under 18 years (20 years in case of Japan) at the time of assent or willingness to participate in the study cannot be confirmed due to MPS I-related intellectual disability, informed permission from the patient's legally acceptable representative (e.g., his/her parents or guardians) need to be obtained instead of his/her consent. Even in this case, written informed consent should be obtained from the patient, wherever possible
* Female patient or male patient whose co-partners is of child-bearing potential agree to use a medically accepted, highly effective method of contraception, such as spermatocidal gel plus condom, an intrauterine device or oral contraceptives until one month after the final administration.

Exclusion Criteria:

* A patient who is unable to perform the study procedures, except for 6-minute walk test, neurocognitive testing, BVMT-R, HVLT-R, and T.O.V.A.
* Judged by the principal investigator or subinvestigator as being unable to undergo lumbar puncture, including those who have difficulties in taking a position for lumbar puncture due to joint contracture or those who are likely to experience difficulty breathing during the lumbar puncture process
* Judged by the principal investigator or subinvestigator to be ineligible to participate in the study due to a history of a serious drug allergy or hypersensitivity to any drugs
* Otherwise judged by the principal investigator or subinvestigator to be ineligible to participate in the study in consideration of patient's safety

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | 156 weeks
  Adverse events
Incidence of abnormal laboratory test results | 156 weeks
  Hematology
Incidence of abnormal laboratory test results | 156 weeks
  Biochemistry
Incidence of abnormal laboratory test results | 156 weeks
  Serum iron tests
Incidence of abnormal laboratory test results | 156 weeks
  Urinalysis
Incidence of abnormal vital signs | 156 weeks
  Pulse rate
Incidence of abnormal vital signs | 156 weeks
  Body temperature
Incidence of abnormal vital signs | 156 weeks
  Blood pressure
Incidence of abnormal vital signs | 156 weeks
  Body weight
Incidence of abnormal EKG readings | 156 weeks
Number of participants with Adverse Events | 156 weeks
  Anti-human-α-L-iduronidase antibodies
Number of participants with Adverse Events | 156 weeks
  Anti-JR-171 antibodies
Number of participants with Adverse Events | 156 weeks
  Infusion associated reaction (IAR)

SECONDARY OUTCOMES:
Change From Baseline in Heparan Sulfate Levels in Cerebrospinal Fluid (CSF) | Weeks 26, 52, 104, 156
Change From Baseline in Dermatan Sulfate Levels in Cerebrospinal Fluid | Weeks 26, 52, 104, 156
CSF opening pressure | Weeks 26, 52, 104, 156
Change From Baseline in Heparan Sulfate Levels in Urinary | Weeks 13, 26, 39, 52, 65, 78, 91, 104, 130, 156
Change From Baseline in Dermatan Sulfate Levels in Urinary | Weeks 13, 26, 39, 52, 65, 78, 91, 104, 130, 156
Change From Baseline in Heparan Sulfate Levels in Serum | Weeks 13, 26, 39, 52, 65, 78, 91, 104, 130, 156
Change From Baseline in Dermatan Sulfate Levels in Serum | Weeks 13, 26, 39, 52, 65, 78, 91, 104, 130, 156
Change From Baseline in Liver Volume | Weeks 13, 26, 52, 78, 104, 156
Change From Baseline in Spleen Volume. | Weeks 13, 26, 52, 78, 104, 156
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  Left ventricular posterior wall thickness
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  interventricular septal thickness
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  left ventricular mass index
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  left ventricular ejection fraction
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  left ventricular ejection fraction,
Change From Baseline in Echocardiography. | Weeks 13, 26, 52, 78, 104, 156
  E/A ratio
Change From Baseline in 6-minute Walk Test Distance. | Weeks 13, 26, 52, 78, 104, 156
Changes from baseline in cognitive age equivalent score of neurocognitive testing | Weeks 52, 104, 156
  Wechsler Intelligence Quotient (IQ) test or the Bayley scales of infant and toddler development
Changes from baseline in outcome of adaptive behavioral function | Weeks 52, 104, 156
  Vineland adaptive behavior scales
Changes from baseline in outcome of the Brief Visuospatial Memory Test-Revised | Weeks 13, 26, 52, 78, 104, 130, 156
Changes from baseline in outcome of the Hopkins Verbal Learning Test-Revised | Weeks 13, 26, 52, 78, 104, 130, 156
Changes from baseline in outcome of the Test of Variables of Attention | Weeks 13, 26, 52, 78, 104, 130, 156
Changes from baseline in outcome of the Pediatric Quality of Life Inventory Family Impact Module (PedsQL-FIM) | Weeks 13, 26, 52, 104 156

CONTACTS AND LOCATIONS:
Locations (6):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Genética e Erros Inatos do Metabolismo - IGEIM, São Paulo
- Japan (3):
  - Fukuoka Children's Hospital, Fukuoka
  - National Hospital Organization Kokura Medical Center, Kitakyushu
  - Osaka Metropolitan University Hospital, Osaka

IPD SHARING:
Plan to Share IPD: No